CLINICAL TRIAL: NCT02200484
Title: Helping Ethnically Diverse Teen Moms Prevent Obesity in Their Preschool Children
Brief Title: Project HERA (Health, Education, and Relationship-building for Adolescents- Moms and Tots)
Acronym: Project HERA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Brown University (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other); University of South Carolina (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14864; R21HL114083 (NIH)
Record Dates: First submitted 2014-07-12; First posted 2014-07-25 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Child Behavior Problems; Parenting Skills; Obesity Prevention
Keywords: obesity; adolescents, females; child development; weight loss programs; child rearing; parenting
MeSH Terms: conditions — Obesity | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Training/Obesity Prevention (Experimental): Mother-child dyads randomized to the active intervention in the pilot study will be administered 8 weeks of a combined parenting training and obesity prevention program that was adapted through analysis of formative research interviews with adolescent mothers with feedback from an expert panel of multidisciplinary research team members and community members.
  Interventions: Behavioral: Combined parent training and obesity prevention program
- 8-week Wellness Program (Control) (Active Comparator): Participants randomized to control condition during intervention piloting will receive print-based health and wellness materials once weekly for 8-weeks + 2 follow up telephone calls at the beginning and conclusion of the 8-week program.
  Interventions: Behavioral: Wellness program (active contact control)

INTERVENTIONS:
Behavioral: Combined parent training and obesity prevention program
  Arms: Parent Training/Obesity Prevention
Behavioral: Wellness program (active contact control)
  Arms: 8-week Wellness Program (Control)

SUMMARY:
Specific Aims:

1. The primary aims of this study are to conduct formative interviews with teen mothers to inform a targeted adaptation of empirically based weight management and parent training programs for teen mothers for their preschoolers.
2. To conduct a small pilot and post-pilot focus group of the feasibility and acceptability of recruitment and retention methods & the intervention.

Study Hypotheses:

Given the small sample size and fact that this is a pilot study, focus will be on estimating effect sizes rather than statistical hypothesis testing. However, the investigators exploratory hypotheses are as follows:

1. (a) The adapted intervention will be more feasible compared to the wellness control condition, with a participant retention rate of ≥80% and an average adherence (attendance at weekly treatment sessions; homework completion 5 weekdays weekly) is ≥ 75%; (b) The adapted intervention will be more acceptable compared to the wellness control condition, based on the Consumer Satisfaction Scale and Therapy Assessment Inventory with ≥90% of the participants responding to the item, "In general how satisfied were you with the intervention?" by choosing "unsatisfied" to "very satisfied."
2. (a) The adapted intervention will result in greater improvements in child behavior and parent-child connectedness compared to the control condition; (b) the adapted intervention versus wellness control condition will result in greater increases in child and teen mother individual as well as joint physical activity and physically active play and greater reductions in individual and joint teen mother and child sedentary behavior (television viewing) from baseline to post-intervention; (c) the greater teen mother and child fruit and vegetable consumption; and reduced child juice and sugar-sweetened beverage consumption from baseline to post-intervention; (d) the adapted intervention versus wellness control condition will result in smaller increases in child BMI percentile and teen mother BMI from baseline to post-intervention; (e) participants who attend higher numbers of intervention sessions will show greater improvements in target outcomes (child behavior, parent-child connectedness, and teen mother and child physical activity, sedentary behavior and BMI); with participants receiving the adapted intervention versus wellness control showing the greatest dose-based improvements.

ELIGIBILITY:
Inclusion Criteria:

* Must be teen moms
* Be between 16 and 20 years of age

Exclusion Criteria:

* Does not have a child between the ages of 6 months and 5 years

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Study Feasibility | Measured at the beginning of participant recruitment through 8 weeks follow up (end of treatment)
  Feasibility will be assessed during intervention piloting using process evaluation data to determine the pace of recruitment relative to sample size goals and differences in retention by condition. Descriptive analyses will determine the % of participants recruited, rate of accrual, attrition rate over time and total, % accepting randomization to treatment, and % compliance with study protocols (as measured by number of sessions attended, number who complete homework, etc…). Due to the small sample size in the current study, the intervention will be considered feasible if the retention rate is ≥ 80% and if the average adherence (attendance at weekly treatment sessions; homework completion 5 weekdays weekly) is ≥ 75%. The post pilot focus group will probe participants about their perspective on methods used to recruitment them into the study, including advertisements, incentives, location etc...
Study Acceptability | 8-weeks follow up (end of treatment)
  We will assess study acceptability via maternal completion of customer satisfaction questionnaires at the end of treatment (8 weeks follow up) for participants randomized (n=46) during intervention piloting to the adapted intervention (combined parenting/obesity prevention program) versus control condition (wellness program). We will invite a subsample of n=8 adolescent mothers to participate in the post-pilot focus group to further assess study acceptability and probe these participants on the likes and dislikes for the program, and recruitment methods.

SECONDARY OUTCOMES:
Change in Child Problem Behavior | Baseline, Each week for 8 weeks during active treatment, and 8-weeks follow up (end of treatment)
  We will assess for changes in child problem behavior via maternal completion of child behavior questionnaires administered at baseline, once weekly for eight weeks during active intervention, and at 8 weeks end of treatment (follow up) for participants randomized (n= 46) to the intervention arm (parenting/combined obesity prevention program) versus control (wellness condition).
Change in Child Physical Activity/Sedentary Behavior | Baseline, 8-weeks follow up (end of treatment)
  Child physical activity and sedentary behavior will be measured via maternal completion of questionnaires administered at baseline and 8 weeks follow up to assess for changes in these outcomes across participants randomized during intervention piloting (n=46) to the intervention condition (combined parenting/obesity prevention program) versus control condition (wellness program). Child physical activity and sedentary behavior will also be assessed via a home audit of the home physical activity/sedentary behavior environment completed by the research assistant at baseline and 8-weeks follow up (end of treatment)
Change in Child fruit, Vegetable, Junk, Fat and Fast food Intake (Child Nutritional Behavior) | Baseline, 8-weeks follow up (end of treatment)
  Child nutritional behavior will be measured via maternal completion of questionnaires administered at baseline and 8 weeks follow up to assess for changes in these outcomes across participants randomized during intervention piloting (n=46) to the adapted intervention condition (combined parenting/obesity prevention program) versus control condition (wellness program). Child nutritional behavior will also be assessed via a home audit completed by the research assistant at baseline and 8-weeks follow up (end of treatment).

OTHER OUTCOMES:
Change in Child Weight Status (BMI percentile) | Baseline, 8-weeks follow up (end of treatment)
  We will measure child height and weight at baseline and 8-weeks follow up (end of treatment) to calculate child BMI percentile to assess for changes in BMI percentile for participants randomized during intervention piloting (n=46) to the adapted intervention condition (combined parenting/obesity prevention program) compared to those in the control condition (wellness program).

CONTACTS AND LOCATIONS:
Locations (1):
- UMass, Worcester, Massachusetts, United States